CLINICAL TRIAL: NCT03097549
Title: Mobile App-treatment of Mixed and Urgency Urinary Incontinence in Women - a Randomized Controlled Study
Brief Title: Mobile App-treatment of Mixed and Urgency Urinary Incontinence in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: Swedish Council for Working Life and Social Research (Other); Jämtland County Council, Sweden (Other Government); Norrlandstingens Regionförbund (Other); Västerbotten County Council, Sweden (Other Government)
Responsible Party: Principal Investigator, Eva Samuelsson, Associate professor, MD, PhD, General Practitioner, Umeå University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Forte 2014-5140
Record Dates: First submitted 2017-03-20; First posted 2017-03-31 (Actual); Results first posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Urinary Incontinence
Keywords: urinary incontinence; urgency urinary incontinence; mixed urinary incontinence; smartphone application; ehealth; mhealth; randomized controlled trial; self management; treatment
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tät®II Treatment app (Experimental): Comprehensive treatment programme with information and exercises. Individual advices.
  Interventions: Device: Tät®II Treatment app
- Tät®II Information app (Other): Information only.
  .
  Interventions: Device: Tät®II Information app

INTERVENTIONS:
Device: Tät®II Information app — Information about pelvic floor muscle training and bladder training for urgency and mixed urinary incontinence. Information about psychological factors and life style factors that might interfere with incontinence.
  Other Names: Mobile application Tät®II with information only
  Arms: Tät®II Information app
Device: Tät®II Treatment app — Information about pelvic floor muscle training and bladder training for urgency and mixed urinary incontinence. Information about psychological factors and life style factors that might interfere with incontinence .Exercises for the pelvic floor muscles, for bladder training, and for behaviours of avoidance due to fear of leakage, a statistic function and possibility to set reminders. Individual advices regarding life style factors and training based on findings from the bladder diary and answers in the questionnaires.
  Other Names: Mobile application Tät®II with treatment programme
  Arms: Tät®II Treatment app

SUMMARY:
The purpose of this study is to determine whether a comprehensive treatment programme for self-management of mixed and urgency urinary incontinence via a mobile app is effective.

DETAILED DESCRIPTION:
Urinary incontinence affects one fourth of adult women (1). It may reduce quality of life and costs for society are high. The most common type in women is stress urinary incontinence (SUI), i.e. leakage when coughing, sneezing or jumping. Urgency urinary incontinence (UUI) and mixed urinary incontinence (MUI), a combination of both stress and urgency UI, together adds up to nearly half of the cases of UI in women (1). Many women do not seek care, sometimes due to embarrassment (2). The recommended first line treatment for all three types of UI in women are pelvic floor muscle training (PFMT) and life style advices, leading to improvement or cure in two thirds of patients (3,4) . In addition, bladder training might be effective for UUI and MUI (3,4). Bladder training in combination with PFMT led to improvement or cure in one sixth of women with MUI (3). Previous research also suggest that psychological treatment could have a value for some women with UUI and MUI (5).

The investigators have previously demonstrated the efficacy of the mobile app Tät® for treatment of SUI (6). Apps have the potential to improve symptoms in many chronic conditions through self-management interventions (7).

The investigators have developed the mobile app Tät®II for women with UUI or MUI and the aim is to determine if this mobile app is effective for self-treatment.

Women are consecutively recruited via the website www.tät.nu (www.econtinence.se). The women answer an online screening questionnaire with automated response for initial screening of eligibility criteria. Informed consent and bladder diary are sent by ordinary post to the administrator of the study. After that, the women answer a web questionnaire including scoring instruments and finally a telephone interview is conducted by a urotherapist or a doctor. The purpose of this telephone interview is to confirm the clinical diagnosis of UUI or MUI, to ascertain that there are no alarm symptoms motivating examination in ordinary health care and to make sure that the woman is well informed about the study procedure.

After the telephone interview it is decided whether the woman is eligible for participation or not. If eligible, the interviewer send an e-mail to the study coordinator marked "Randomization". The order in which these e-mails arrive at the incoming mail box tat2.am@umu.se decide the order of randomization. An independent administrator has generated the allocation sequence and prepared 130 numbered opaque sealed envelopes (with assignment equally distributed between the two study groups). The study coordinator consecutively opens one envelope for each participant (in the order they arrived in the mailbox) and mark the number of the envelope on the coordinator list for the participant. The coordinator assigns an e-mail to the participant, with instructions for downloading the apps. If assigned to the treatment app group, a unique code is activated for each participant, which enables the participant to activate the complete app Tät®II including individual advices regarding self-care and recommended exercises based on the results from the questionnaire and the bladder diary. Two weeks after randomization, the activation status of the app is controlled and if it is not activated, the participants receive an e-mail asking whether they have experienced any technical problems with the app. In case of technical problems, they get instructions by e-mail or by telephone. After another week, a new review of the activation status is done and if the app still is not activated - participants are contacted via telephone.

Adverse events All participants are encouraged to report any adverse events that may occur during the study either by e-mail or by telephone. This information is included in the e-mail they get after allocation to treatment app or information app group. Questions about adverse events are also included in the follow-up questionnaire

14 weeks after randomization, the study coordinator will send both groups a web-based questionnaire with follow-up questions and scoring instruments and a bladder diary. The bladder diary is sent back by post. Non-responders will be reminded twice by e-mail (at 2 and 4 weeks) and once by telephone (at 6 weeks).

The participants in the information app group will receive an unique activating code to get access to the complete app with individual advices after this follow-up. The participants in the original information app group will be followed-up after another 14 weeks with the same follow-up questionnaire and a bladder diary and the same time frames for reminders. The results from this second follow-up in the original information app group will be compared with results from the first follow-up and serve as quality control for the original study. This design allows us to study long-term follow up results later.

Quality Assurance plan The study will be monitored according to Good Clinical Practice principles by study research nurse Agneta Lindberg at the local Clinical Research Centre of Region Jämtland Härjedalen to ascertain a proper procedure of conduction, recording and reporting data. The monitor will review study records, observe protocol procedures and the randomization process, and ensure that written informed consent has been correctly obtained. The first five participants-and after that one in ten randomly selected by the monitor- will be 100 % monitored as stated in the monitor plan. All study participants will be reviewed for informed consent procedure. According to the Medical Devices Directives (Meddevs 2.7/3) reporting and monitoring of adverse events and serious adverse events are not necessary when a CE-marked (Conformité Européenne) device is used in a study within its intended use covered by the CE-marking. The app Tät®II is used within its intended use covered by the CE-marking (Medical Product Agency, Sweden. Dnr:6.6.1-2016-97327, PID (Product identify number) 149104).

Data Dictionary, see primary and secondary outcomes

Plan for missing data The questionnaires will be web-based and every question will, if technically possible, be mandatory. However, should there for some reason be missing values, these will be replaced with the value corresponding to "no change", i.e. a missing value at follow-up will be replaced with the participant´s baseline value and a missing value at baseline will be replaced with the follow-up value. A missing answer in the PGI-I at follow-up will be assumed as "unchanged".

All data will be checked for out-of-range results, these will be treated as missing values.

Sample size calculation Based on results from the previous smartphone study and the findings of Albers-Heitner et al, improvements in the ICIQ UI SF of 2.5 points in the treatment app group and 0.9 points in the information app group are assumed. To detect this difference with 80% power, 2-side test and significance 0.05, a sample size of 49 is needed in each group. With an expected drop-out rate of 20%, approximately 60 participants are needed in each group. The investigators therefore aim to recruit 120 women aged 18 and older via the website www.tät.nu.

Statistical plan Intention-to-treat analysis will be performed on all outcome measures.

Baseline The two groups will be compared at baseline using Student´s t-test for continuous variables, Pearson Chi-Square test for categorical variables, and the Mann-Whitney U-test for ordinal variables. Baseline data will be compared for age, BMI, educational level, medication and for all primary and secondary outcomes that are measured at baseline.

Primary outcome The primary outcome is the difference between the groups in mean ICIQ UI SF score at follow-up and a linear mixed model analysis incorporating baseline data will be used.

Secondary outcomes

Comparison between groups:

For evaluating the difference between the groups in mean ICIQ LUTS qol score at follow-up, a linear mixed models analysis incorporating baseline data will be used.

For evaluating the difference between the groups regarding change of the median Incontinence Episode Frequency from baseline to follow-up, the Mann-Whitney U-test will be used.

To evaluate the difference between the groups in mean ICIQ-OAB score at follow-up, a linear mixed models analysis will be used incorporating baseline data.

To evaluate the difference between the groups in the mean score of the non-validated Incontinence Catastrophizing Scale (ICS) at follow-up, a linear mixed models analysis will be used incorporating baseline data.

For evaluating the difference between groups regarding change in usage of incontinence aids from baseline to follow-up, the Mann-Whitney U-test will be used.

The difference between the groups regarding PGI-I, a question on improvement only used at follow-up, will be analysed using the Mann-Whitney U-test.

Patient satisfaction. The proportion of participants that intend to seek more help after this first-line treatment will be analysed, this item will only be analysed in the treatment app group and no comparisons will be done.

Comparison within groups:

For comparison within the groups regarding the score on ICIQ LUTS qol, a paired t-test will be used.

For comparison within the groups regarding the IEF, a Wilcoxon signed-rank test will be used.

For comparison within the groups regarding the score on ICS, a paired t-test will be used For comparison within the groups regarding the score on ICIQ-OAB, a paired t-test will be used.

For comparison within the groups regarding the incontinence aid usage, a Wilcoxon signed-rank test will be used.

ELIGIBILITY:
Inclusion Criteria:

* Urgency urinary incontinence or mixed urinary incontinence, established via telephone interview
* Urinary leakage twice a week or more often
* Duration of urinary leakage with urgency for at least 12 months
* Ability to read and write Swedish
* Asset to a smartphone (minimum iOS* 8.0 for Apple, 4.0.3 for Androids
* Possibility to send and receive email and asset to printer
* Motivation and time to perform a 15 weeks long treatment programme with focus on self-care and behavioural training (mainly pelvic floor muscle training and bladder training).
* Accept to be randomized to one of two groups; a treatment app group or an information app Group

  * iOS=mobile operating system including iPhone, iPad and iPod touch

Exclusion Criteria:

* Participation in our previous internet or smartphone study
* Ongoing pregnancy
* Former incontinence surgery
* Known malignancy in lower abdomen
* Unassessed difficulties in emptying bladder
* Visual blood in urine
* Three or more urinary tract infections during the last 12 months
* One or more pyelonephritis during the last three years
* Painful micturition
* Painful urgency
* Intermenstrual bleeding
* Neurological disease such as multiple sclerosis or Parkinsons disease
* Previous stroke
* Diabetes mellitus
* Maximum voided volume of less than 150 ml (micturition chart)
* Regular use of any mobile app for pelvic floor muscle training during the last month
* Usage of antimuscarinic drugs or mirabegron during the last month

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2017-04-03 (Actual); Primary Completion 2018-07-27 (Actual); Study Completion 2018-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eva C Samuelsson, MD, PhD, Principal Investigator — Department of public health and clinical medicine, Umeå university, Umeå, Sweden
Locations (1):
- Umea University, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hannestad YS, Rortveit G, Sandvik H, Hunskaar S; Norwegian EPINCONT study. Epidemiology of Incontinence in the County of Nord-Trondelag. A community-based epidemiological survey of female urinary incontinence: the Norwegian EPINCONT study. Epidemiology of Incontinence in the County of Nord-Trondelag. J Clin Epidemiol. 2000 Nov;53(11):1150-7. doi: 10.1016/s0895-4356(00)00232-8. PMID 11106889
- [Background] Siddiqui NY, Levin PJ, Phadtare A, Pietrobon R, Ammarell N. Perceptions about female urinary incontinence: a systematic review. Int Urogynecol J. 2014 Jul;25(7):863-71. doi: 10.1007/s00192-013-2276-7. Epub 2013 Dec 6. PMID 24310988
- [Background] Shamliyan T, Wyman J, Kane RL. Nonsurgical Treatments for Urinary Incontinence in Adult Women: Diagnosis and Comparative Effectiveness [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2012 Apr. Report No.: 11(12)-EHC074-EF. Available from http://www.ncbi.nlm.nih.gov/books/NBK92960/ PMID 22624162
- [Background] Dumoulin C, Hunter KF, Moore K, Bradley CS, Burgio KL, Hagen S, Imamura M, Thakar R, Williams K, Chambers T. Conservative management for female urinary incontinence and pelvic organ prolapse review 2013: Summary of the 5th International Consultation on Incontinence. Neurourol Urodyn. 2016 Jan;35(1):15-20. doi: 10.1002/nau.22677. Epub 2014 Nov 15. PMID 25400065
- [Background] Garley A, Unwin J. A case series to pilot cognitive behaviour therapy for women with urinary incontinence. Br J Health Psychol. 2006 Sep;11(Pt 3):373-86. doi: 10.1348/135910705X53876. PMID 16870050
- [Background] Asklund I, Nystrom E, Sjostrom M, Umefjord G, Stenlund H, Samuelsson E. Mobile app for treatment of stress urinary incontinence: A randomized controlled trial. Neurourol Urodyn. 2017 Jun;36(5):1369-1376. doi: 10.1002/nau.23116. Epub 2016 Sep 9. PMID 27611958
- [Background] Whitehead L, Seaton P. The Effectiveness of Self-Management Mobile Phone and Tablet Apps in Long-term Condition Management: A Systematic Review. J Med Internet Res. 2016 May 16;18(5):e97. doi: 10.2196/jmir.4883. PMID 27185295
- [Background] Albers-Heitner PC, Lagro-Janssen TA, Joore MM, Berghmans BL, Nieman FF, Venema PP, Severens JJ, Winkens RR. Effectiveness of involving a nurse specialist for patients with urinary incontinence in primary care: results of a pragmatic multicentre randomised controlled trial. Int J Clin Pract. 2011 Jun;65(6):705-12. doi: 10.1111/j.1742-1241.2011.02652.x. PMID 21564445
- [Derived] Funada S, Yoshioka T, Luo Y, Sato A, Akamatsu S, Watanabe N. Bladder training for treating overactive bladder in adults. Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD013571. doi: 10.1002/14651858.CD013571.pub2. PMID 37811598
- [Derived] Wadensten T, Nystrom E, Franzen K, Lindam A, Wasteson E, Samuelsson E. A Mobile App for Self-management of Urgency and Mixed Urinary Incontinence in Women: Randomized Controlled Trial. J Med Internet Res. 2021 Apr 5;23(4):e19439. doi: 10.2196/19439. PMID 33818395
- See also: website with information and registration for the study (www.econtinence.se). — http://econtinence.se/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After enrollment, each respondent was contacted via telephone by a specialist incontinence nurse or general practitioner. A telephone interview was conducted with the objectives of confirming the symptom diagnosis (ie, UUI or MUI), reconfirming the absence of exclusion criteria, and ensuring that the participant was fully informed about the study. Of the 142 enrolled,19 participants were found ineligible at the telephone interview.
Groups:
- Tät®II Treatment App: Comprehensive treatment programme with information and exercises. Tailored advice.
  Tät®II Treatment app: Information about pelvic floor muscle training and bladder training for urgency and mixed urinary incontinence. Information about psychological factors and life style factors that might interfere with incontinence .Exercises for the pelvic floor muscles, for bladder training, and for behaviours of avoidance due to fear of leakage, a statistic function and possibility to set reminders. Automated feedback. Tailored advice regarding life style factors and training based on findings from the bladder diary and answers in the questionnaires.
- Tät®II Information App: Information only.
  .
  Tät®II Information app: Brief information about pelvic floor muscle training and bladder training for urgency and mixed urinary incontinence. Brief information about psychological factors and life style factors that might interfere with incontinence.
Period: Overall Study
Arm/Group | Tät®II Treatment App | Tät®II Information App
Started | 60 | 63
Completed | 58 | 63
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tät®II Treatment App | Tät®II Information App | Total
Number analyzed (Participants) | 60 | 63 | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (9.2) | 57.7 (9.9) | 58.3 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Only women were included in the study.
  Participants
    Female | 60 | 63 | 123
    Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: kg/m2] | 26.5 (3.6) | 25.9 (5.2) | 26.2 (4.5)
University education >=3 years, n (%) [Count of Participants; unit: Participants] | 44 | 35 | 79
Self-rated knowledge in using computers or tablets (1-4 points) [Mean (Standard Deviation); unit: units on a scale] — A one-item question about self-perceived knowledgeability when using computers and tablets (4 response options, ranging from "not at all knowledgeable" to "very knowledgeable"). Range 0-4 points, higher score indicating greater knowledgeability. This question was derived from the 2016 Swedish national survey "Svenskarna och Internet" (The Swedes and the Internet).
  units on a scale | 3.5 (0.6) | 3.4 (0.6) | 3.4 (0.6)
eHEALS score [Mean (Standard Deviation); unit: units on a scale] — Measures e-Health literacy and digital competence. eHEALS = The eHealth Literacy Scale. Includes 8 items. Total score ranges from 8-40 points. Higher scores indicate a higher level of eHealth literacy.
  units on a scale | 32.85 (5.59) | 33.83 (4.51) | 33.35 (5.07)
Physical activity >3 hours/week [Count of Participants; unit: Participants] | 33 | 40 | 73
Smoker [Count of Participants; unit: Participants] | 1 | 2 | 3
Coffee consumption >= 5 cups/day [Count of Participants; unit: Participants] | 7 | 10 | 17
Tea consumption >= 5 cups/day [Count of Participants; unit: Participants] | 4 | 2 | 6
Often or always constipated [Count of Participants; unit: Participants] | 6 | 3 | 9
Never given birth [Count of Participants; unit: Participants] | 8 | 7 | 15
Postmenopausal >1 year [Count of Participants; unit: Participants] | 42 | 47 | 89
Local estrogen usage [Count of Participants; unit: Participants] | 11 | 13 | 24
Systemic estrogen usage [Count of Participants; unit: Participants] | 1 | 1 | 2
Hysterectomy [Count of Participants; unit: Participants] | 4 | 7 | 11
Prolapse surgery [Count of Participants; unit: Participants] | 3 | 0 | 3
Incontinence surgery [Count of Participants; unit: Participants] | 3 | 3 | 6
Mixed urinary incontinence [Count of Participants; unit: Participants] | 45 | 43 | 88
Urgency urinary incontinence [Count of Participants; unit: Participants] | 15 | 20 | 35
Duration of urinary incontinence symptoms >5 years [Count of Participants; unit: Participants] | 37 | 38 | 75
Previous health care contact for incontinence symptoms [Count of Participants; unit: Participants] | 19 | 19 | 38
ICIQ-UI SF score [Mean (Standard Deviation); unit: units on a scale] | 11.71 (3.48) | 11.44 (3.20) | 11.58 (3.33)
IEF per week [Mean (Standard Deviation); unit: urinary leakage episodes/week] | 21.82 (16.80) | 21.06 (13.71) | 21.43 (15.23)

OUTCOME MEASURES:

1. Primary Outcome: International Consultation on Incontinence Modular Questionnaire Urinary Incontinence Short Form (ICIQ-UI SF)
Description: Three items on frequency, amount of leakage and overall impact. Scoring 0-21, higher values indicating increasing severity.
Time Frame: 15 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tät®II Treatment App | Tät®II Information App
Number analyzed (Participants) | 58 | 63
score on a scale | 7.0 (3.7) | 9.8 (3.5)
Statistical Analysis 1: Comparison: Tät®II Treatment App vs Tät®II Information App; Comparison of mean scores using a linear mixed model, incorporating baseline data and accounting for all available data. Sample size calculation: We anticipated ICIQ-UI SF improvements of 2.5 points in the treatment group and 0.9 points in the information group. Detecting this difference with 80% power, a two-sided test, and a significance level of P<.05 would require a sample size of 49 in each group. With an expected drop-out rate of 20%, we needed approximately 60 participants in each group; Test type: Superiority; p = 0.001, Mixed Models Analysis; Estimated difference = -3.1, 95% CI 2-sided [-4.8 to -1.3]

2. Secondary Outcome: International Consultation on Incontinence Modular Questionnaire Lower Urinary Tract Symptoms Quality of Life (ICIQ- LUTSqol).
Description: The instrument includes 19 items on the impact of the leakage. All items are scored 1-4 (not at all/never, slightly/sometimes, moderately/often, a lot/all the time). The overall score is 19-76, with higher values indicating increased impact on QOL.
Time Frame: 15 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tät®II Treatment App | Tät®II Information App
Number analyzed (Participants) | 58 | 63
score on a scale | 29.8 (7.8) | 36.5 (9.0)
Statistical Analysis 1: Comparison: Tät®II Treatment App vs Tät®II Information App; Null hypothesis: There is no difference in score between the treatment group and the information group at follow-up; Test type: Superiority; p = 0.004, Mixed Models Analysis; Estimated difference = -6.3, 95% CI 2-sided [-10.5 to -2.1]

3. Secondary Outcome: Change From Baseline Incontinence Episode Frequency (IEF)
Description: Number of incontinence episodes per 48 hours transferred to per week.
Time Frame: 15 weeks
Measure: Median (Inter-Quartile Range); unit: urinary leakage episodes/week
Arm/Group | Tät®II Treatment App | Tät®II Information App
Number analyzed (Participants) | 60 | 63
urinary leakage episodes/week | 3.5 [0.0 to 10.5] | 10.5 [7.0 to 21.0]
Statistical Analysis 1: Comparison: Tät®II Treatment App vs Tät®II Information App; Null hypothesis: There is no difference in the number of urinary leakage episodes between the treatment app users and the information app users at follow-up. ITT analysis. Missing data: 5 participants in the treatment group and 2 participants in the information group had a missing value at follow-up, and for those, the difference was set to 0 (ie, no change); Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: International Consultation on Incontinence Modular Questionnaire Overactive Bladder (ICIQ-OAB)
Description: Four items on frequency of micturition during day and during night, frequency of urgency and urgency leakage, each item scored 0-4, total score 0-16, higher values indicating increased severity.
Time Frame: 15 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tät®II Treatment App | Tät®II Information App
Number analyzed (Participants) | 58 | 63
score on a scale | 4.7 (2.0) | 6.4 (2.0)
Statistical Analysis 1: Comparison: Tät®II Treatment App vs Tät®II Information App; Null hypothesis: There is no difference in score between the treatment group and the information group at follow-up; Test type: Superiority; p < 0.001, Mixed Models Analysis; Estimated difference = -1.8, 95% CI 2-sided [-2.8 to -0.9]

5. Secondary Outcome: Incontinence Catastrophizing Scale (ICS)
Description: Seven items on fear of leakage and urgency. Alternatives on each item; Never (=0), sometimes (=1), often (=2), Always (=3). Score 0-21.
Time Frame: 15 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tät®II Treatment App | Tät®II Information App
Number analyzed (Participants) | 58 | 63
score on a scale | 2.3 (2.1) | 4.1 (2.5)
Statistical Analysis 1: Comparison: Tät®II Treatment App vs Tät®II Information App; Null hypothesis: There is no difference in score between the treatment group and the information group at follow-up; Test type: Superiority; p = 0.016, Mixed Models Analysis; Estimated difference = -1.6, 95% CI 2-sided [-2.8 to -0.3]

6. Secondary Outcome: Change From Baseline Usage of Incontinence Aids at 15 Weeks
Description: Use of incontinence aids during the last four weeks, six response options from "Never" to "more than one incontinence aid per day"
Time Frame: 15 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Tät®II Treatment App | Tät®II Information App
Number analyzed (Participants) | 58 | 63
Participants
  Less than once a week | 38 | 25
  Once a week or more | 20 | 38
Statistical Analysis 1: Comparison: Tät®II Treatment App vs Tät®II Information App; Null hypothesis: no difference in usage between treatment group and information group at follow-up; Test type: Superiority; p = 0.01, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Patient Global Impression of Improvement (PGI-I)
Description: Validated 7-item scale on improvement from very much improved to very much worse.
Time Frame: 15 weeks
Population: Missing values for two participants in the treatment group were imputed as "no change".
Measure: Count of Participants; unit: Participants
Arm/Group | Tät®II Treatment App | Tät®II Information App
Number analyzed (Participants) | 60 | 63
Participants
  Any improvement | 52 | 19
  No change, or worsened condition | 8 | 44
Statistical Analysis 1: Comparison: Tät®II Treatment App vs Tät®II Information App; Null hypothesis: No difference in improvement between the treatment group and the information group att follow-up; Test type: Superiority; p < 0.001, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Patient Satisfaction
Description: A self-rated question about if the current treatment was sufficient, with three response options.
Time Frame: 15 weeks, only for the Tät® II treatment app group
Population: Missing values for 5 participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Tät®II Treatment App
Number analyzed (Participants) | 55
Participants
  Satisfied with the treatment | 35
  Not satisfied, but not considering seeking additional care | 13
  Not satisfied, and considering seeking additional care | 7

ADVERSE EVENTS:
Time Frame: Treatment app group:15 weeks from randomisation. Information app group: 15 weeks from randomisation
Description: Participants were informed to contact the study team in case of any adverse events during the study via e-mail or via telephone.
Arm/Group | Tät®II Treatment App | Tät®II Information App
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/63
Other Adverse Events (participants affected / at risk) | 2/60 | 0/63
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tät®II Treatment App (N=60) | Tät®II Information App (N=63)
Inguinal hernia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — One participant reported the development of an inguinal hernia during the treatment period, which later required surgery. Discussion of this case with specialists led to the conclusion that the hernia was likely not related with the use of the app.
Altered incontinence symptoms (Renal and urinary disorders) | 1 (1) | 0 (0) — One participant reported altered incontinence symptoms, with decreased urgency but increased episodes of spontaneous urinary leakage.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-04): https://cdn.clinicaltrials.gov/large-docs/49/NCT03097549/Prot_SAP_000.pdf